CLINICAL TRIAL: NCT03290014
Title: Sleep Quality in COPD Patients. A Clinical and Polysomnographic Study
Brief Title: Sleep Quality in (COPD) Patients (COPD: Chronic Obstructive Pulmonary Disease)
Acronym: COPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: PR(AG)365/2015
Record Dates: First submitted 2017-09-08; First posted 2017-09-21 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-09

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Polysomnography; Actigraphy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Good sleepers: COPD patients with good sleep quality according to CASIS score will be studied with polysomnography, actigraphy and OSLER test
  Interventions: Diagnostic Test: polysomnography; Diagnostic Test: Actigraphy; Diagnostic Test: Osler test
- Bad sleepers: COPD patients with poor sleep quality according to CASIS score will be studied with polysomnography, actigraphy and OSLER test
  Interventions: Diagnostic Test: polysomnography; Diagnostic Test: Actigraphy; Diagnostic Test: Osler test

INTERVENTIONS:
Diagnostic Test: polysomnography — Monitoring of brain activity and respiratory variables during sleep
Diagnostic Test: Actigraphy — monitoring daily physical activity for 7 days
Diagnostic Test: Osler test — Evaluation of subjects´ ability to remain awake
  Other Names: Oxford sleep resistance test

SUMMARY:
Patients with COPD, in addition to daytime symptoms, may suffer from nocturnal disturbances. The frequency of nocturnal problems has been reported to be higher in COPD than in the general population and it currently affects up to 50% of patients.

The CASIS questionnaire includes 7 questions and it has been recently validated as an objective tool to evaluate nocturnal symptoms in patients with asthma and COPD. The present study aims to study the validity of the CASIS questionnaire as a predictor of sleep quality measured by objective polysomnographic parameters.

ELIGIBILITY:
Inclusion criteria:

Patients with written inform consent to participate in the study and all the following criteria will be selected:

* Age 40-80 years
* Smokers or exsmokers of at least 10 pack-years
* Moderate-to-severe COPD

Exclusion criteria:

* Non-stable COPD. Stability is defined as being exacerbation free and without treatment changes for at least 4 weeks prior to baseline evaluation. The presence of a COPD exacerbation previous to the sleep studies (polysomnography, actigraphy, OSLER test) will lead to an early discontinuation of the patient´s participation in the study.
* Heart failure, asthma, cancer or other major medical illness with known effects on sleep quality.
* Unable to understanding the questionnaires administered in the study.
* Known Obstructive Sleep Apnea, other sleep disorder (narcolepsy, periodic limb movements) or shift work.
* Chronic respiratory failure (PaO2 <60 mmHg).
* Treatment with sedatives or antidepressants.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients aged 40-80 years, smokers or exsmokers of at least 10 pack-years, diagnosed with moderate-to-severe COPD (post bronchodilator FEV1% < 70% and FEV1 ≥ 30 but < 80% of predicted in a spirometry performed within 6 months prior to inclusion into the study)
Sampling Method: Non-Probability Sample
Enrollment: 58 (Estimated)
Dates: Start 2017-03-01 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-09-30 (Estimated)

PRIMARY OUTCOMES:
Sleep efficiency | One night at the sleep unit
  Sleep time/Time in bed

SECONDARY OUTCOMES:
Total sleep time | One night at the sleep unit
  Total sleep time
Arousal index | One night at the sleep unit
  number of arousals/hour of sleep
sleep architecture | One night at the sleep unit
  percentage of the different sleep phases
Osler test error index | Next morning after polysomnography (8a.m.--4 p.m.)
  number of errors
Actigraphy | One week previous to polysomnography
  Monitoring of rest/activity cycles

CONTACTS AND LOCATIONS:
Overall Officials: Marc Miravitlles, PhD, Study Chair — Vall d´Hebron Institut de Recerca
Locations (1):
- Hospital Universitari Vall d´Hebron, Barcelona, Spain

REFERENCES:
- [Background] Pokrzywinski RF, Meads DM, McKenna SP, Glendenning GA, Revicki DA. Development and psychometric assessment of the COPD and Asthma Sleep Impact Scale (CASIS). Health Qual Life Outcomes. 2009 Dec 7;7:98. doi: 10.1186/1477-7525-7-98. PMID 19968881
- [Background] Miravitlles M, Iriberri M, Barrueco M, Lleonart M, Villarrubia E, Galera J. Usefulness of the LCOPD, CAFS and CASIS scales in understanding the impact of COPD on patients. Respiration. 2013;86(3):190-200. doi: 10.1159/000341175. Epub 2012 Oct 2. PMID 23037958

DOCUMENTS (1):
  • Study Protocol (2016-06-10): https://cdn.clinicaltrials.gov/large-docs/14/NCT03290014/Prot_000.pdf